CLINICAL TRIAL: NCT05169697
Title: A Multicenter, Open-label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of YH002 in Combination with YH001 in Subjects with Advanced Solid Tumors
Brief Title: A Study to Assess YH002 in Combination with YH001 in Subjects with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH002004
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- YH002 in combination with YH001 (Experimental): Dose escalation:A traditional 3+3 dose escalation algorithm will be utilized to identify MTD and/or RP2D Dose expansion:One selected dose after the escalation stage will be expanded to enroll additional 20 subjects. The subjects will be divided into two groups：A and B.
  Interventions: Drug: A:YH002+YH001; Drug: B:YH002+YH001; Drug: YH002+YH001

INTERVENTIONS:
Drug: A:YH002+YH001 — YH002 on CnD1,YH001 on CnD8,Q3W
Drug: B:YH002+YH001 — YH002 and YH001 on same day,Q3W
Drug: YH002+YH001 — A traditional 3+3 dose escalation algorithm

SUMMARY:
A multicenter, open-label, phase I dose escalation study to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of YH002 in combination with YH001 in subjects with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry patients must satisfy all of the following criteria:

1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
2. Subjects must have histologically advanced or cytologically confirmed solid tumor and and must have at least 1 unidimensional measurable lesion by RECIST 1.1.
3. Subjects have progressed on after treatment with at least one standard therapy, or intolerant of the standard therapy, or no standard therapy accessible to the patients due to any reason.
4. Subjects must be age 18 to 80 years of age at the time of screening.
5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥3 months based on investigator's judgement.
7. Subjects have adequate bone marrow and other organ function at the screening visit.
8. Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test within 7 days of the first dosing. Women of reproductive potential are those who have not been post-menopausal for at least 12 months or who have not undergone bilateral tubal occlusion, hysterectomy, or bilateral salpingectomy.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be enrolled:

1. Subjects have another active invasive malignancy within 5 years.
2. Previous exposure to TNFR such as anti-OX40 antibodies.
3. Subjects must not have received any anticancer therapy or another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of the study treatment(subject to the longer one).
4. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that have not recovered to ≤ Grade 1 per CTCAE 5.0, except alopecia ≤ Grade 2.
5. Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.
6. Subjects must not have a known or suspected history of an autoimmune disorder, including but not limited to inflammatory bowel disease, celiac disease, Wegner syndrome, Hashimoto syndrome, systemic lupus erythematosus, scleroderma, sarcoidosis, or autoimmune hepatitis, within 3 years of the first dose of study treatment.
7. Clinically uncontrolled intercurrent illness, including but not limit to an ongoing active infection, active coagulopathy, uncontrolled diabetes (blood glucose > 250 mg/dl), uncontrolled pleural and peritoneal effusion, psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies
8. Subjects must not have active infection of human immunodeficiency virus, hepatitis B, hepatitis C or Covid-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Determined the maximum tolerated dose (MTD) | Up to 1 year after the last dosing
  The safety profile of combination treatment will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
Determined the recommended Phase II dose (RP2D) | Up to 1 year after the last dosing
  The safety profile of combination treatment will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hongming Pan, Principal Investigator — Sir Run Run Shaw Hospital
Locations (9):
- Australia (4):
  - Orange Health Services, Orange, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
- China (5):
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No